CLINICAL TRIAL: NCT03273309
Title: Comparison of Vibratory Perineal Stimulus With Transvaginal Electrical Stimulation in Women With Urinary Incontinence: a Randomized Clinical Trial
Brief Title: Comparison of Vibratory Perineal Stimulus With Transvaginal Electrical Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16-0064
Record Dates: First submitted 2017-07-26; First posted 2017-09-06 (Actual); Last update posted 2018-03-12 (Actual); Status verified 2017-08

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vibratory Perineal Stimulus (Active Comparator): It's thought that the vibratory perineal stimulation can produces afferent nerve impulses that goes to the sacral spinal cord (S2-S4) via the pudendal nerve and stimulates the sacral somatic response which will cause the pelvic muscle contraction.
  Interventions: Other: Vibratory Perineal Stimulus
- Transvaginal Electrical Stimulation (Active Comparator): Transvaginal electrical stimulation can produces direct and reflex responses of the pelvic floor muscles, being more effective in patients who can't voluntarily contract this musculature. In addition, it increases blood flow to the muscles, restores neuromuscular connections and improves muscle fiber function.
  Interventions: Other: Transvaginal Electrical Stimulation

INTERVENTIONS:
Other: Vibratory Perineal Stimulus — Vibratory perineal stimulus will be applied in patients randomized to this group through an intravaginal probe which emits vibratory pulses, with the device fixed in the following parameters:on time = 8 seconds, off time = 16 seconds, total time = 20 minutes. The intervention time will be 6 weeks, with sessions held once a week.
  Arms: Vibratory Perineal Stimulus
Other: Transvaginal Electrical Stimulation — The transvaginal electrical stimulation will be applied in patients randomized to this group through an intravaginal probe which emits electrical pulses, with the device fixed in the following parameters: frequency = 50 Hz, pulse width = 300ms,on time = 8 seconds, off time = 16 seconds, total time = 20 minutes. The intervention time will be 6 weeks, with sessions held once a week.
  Arms: Transvaginal Electrical Stimulation

SUMMARY:
Aim: To compare the effects of Vibratory Perineal Stimulus with transvaginal electrical stimulation to the pelvic floor muscles functionality in women with urinary incontinence and who are unable to voluntarily contract their pelvic floor muscles.

Study Design: Randomized controlled trial

DETAILED DESCRIPTION:
* The purpose of this study is to find out the effect of vibratory perineal stimulus compared to transvaginal electrical stimulation on the functionality of pelvic floor muscles in women with urinary incontinence who are unable to perform voluntary contraction of this musculature.
* Study Design: Randomized controlled trial
* Search location: The data will collected at the Ambulatory of Urogynecology and Obstetrics of Porto Alegre Clinical Hospital (HCPA), where the activities of Pelvic Physiotherapy are performed.and in the Clinical Research Center of the same hospital.
* Inclusion criteria: women with urinary incontinence with zero or one strength degree of pelvic floor muscle contraction by the Modified Oxford Scale.
* Main outcome: Improvement the functionality of pelvic floor muscles
* Secondary outcome: Improvement of urinary loss
* First protocol: patients will be referred by the medical team and will undergo physiotherapeutic evaluation to collect personal data, check the symptoms of urinary incontinence, apply a quality of life questionnaire and measure pelvic floor muscles strength. If patient has zero or one degree of pelvic floor muscle strength, will be referred to the second phase.
* Second protocol: Patients will be randomized into two groups - Vibratory stimulus group or electrical stimulation group. Both will follow a 6-week treatment protocol with intervention once a week. Both are intravaginal devices applied for 20 minutes, with on cycle of 8 seconds and off cycle of 16 seconds.
* Final protocol: patients will repeat the initial evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of urinary incontinence;
* To be unable to perform a voluntarily contraction of pelvic floor muscles;
* Understand the instruments used in the research;

Exclusion Criteria:

* Allergy to latex;
* Individual or group pelvic floor muscle training in the last 6 months.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2017-11-15 (Actual); Study Completion 2017-11-15 (Actual)

PRIMARY OUTCOMES:
Improvement in pelvic floor muscles functionality | six weeks
  Will be assessed by the PERFECT scheme. Each letter that compose the word means a condition to be evaluated: P = power, E = endurance, R = repetitions, F = fast contractions, E = elevation, C=co-contraction, T= cough reflex.

SECONDARY OUTCOMES:
Improvement of urinary Incontinence | six weeks
  ICIQ-SF - "International Consultation on Incontinence Questionnaire - Short Form". This questionnaire assesses the type of urinary loss, intensity and impact on quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: José Geraldo F Lopes Ramos, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Brazil

IPD SHARING:
Plan to Share IPD: Undecided